CLINICAL TRIAL: NCT01305902
Title: Substance Use and Fitness: A Pilot Study of Contingency Management in Older Adults
Brief Title: Substance Use and Fitness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-040-2; P30DA023918 (NIH)
Record Dates: First submitted 2011-02-25; First posted 2011-03-01 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Substance Abuse; Exercise
MeSH Terms: conditions — Substance-Related Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- walking recommendations (No Intervention): Participants assigned to this condition will be instructed to wear a pedometer daily and scheduled for weekly meetings over for the next 12 weeks. Each week, they will be congratulated if they walked the target goal on any days, and encouraged to meet the goals for the upcoming week. However, they will not receive any tangible reinforcement for walking. The meetings will be brief (about 15 minutes) and will include discussions and handouts related to the health benefits of walking.
- contingency management for walking (Experimental): Participants assigned to this condition will be asked to wear a pedometer daily and scheduled for weekly meetings over for the next 12 weeks. The meeting duration and structure will be similar to that in the standard treatment condition including the handouts, with one exception. Participants in this condition will earn tangible reinforcement in the form of prizes for walking the target number of steps per day.
  Interventions: Behavioral: contingency management

INTERVENTIONS:
Behavioral: contingency management — Participants assigned to the experimental group will earn chances to win prizes if they have walked the recommended number of steps.
  Arms: contingency management for walking

SUMMARY:
The purpose of this pilot study is to estimate the effect size of a contingency management procedure that reinforces walking at rates consistent with the American College of Sports Medicine recommendations of 10,000 or more steps per day in older adults. We expect that participants randomized to the contingency management intervention will increase walking to a greater degree than those assigned to a standard care condition.

ELIGIBILITY:
Inclusion Criteria:

* age 55 - 75 years
* currently not physically active
* willing and physically able as determined by physician approval to walk 10,000 steps per day
* blood pressure of 120-159 mmHg systolic or 80-99 mmHg diastolic
* willing to meet with research staff weekly for 12 weeks

Exclusion Criteria:

* psychiatric or physical illness that could interfere with participation

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
number of days on which participants walked the recommended number of steps | Weeks 1-12

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Petry, Ph.D., Principal Investigator — University of Conncecticut Health Center
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States